CLINICAL TRIAL: NCT00001520
Title: The Early Reversibility of Rocuronium After Different Doses of Neostigmine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 960122; 96-CC-0122
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-09

CONDITIONS: Paralysis
Keywords: Endotracheal Intubation; Neuromuscular Blockade; Neuromuscular Blocking Agents; Paralysis; Reversal Agents
MeSH Terms: conditions — Paralysis | interventions — Neostigmine

INTERVENTIONS:
Drug: neostigmine

SUMMARY:
Neuromuscular blocking agents are commonly used to facilitate endotracheal intubation. Succinylcholine, an ultra short-acting, depolarizing neuromuscular blocking agent, is the most commonly used agent for paralysis in this setting because of its rapid onset and short duration of paralysis. In patients with contraindications to succinylcholine or in whom a difficult airway is anticipated, a neuromuscular blocking agent with a pharmacodynamic profile similar to succinylcholine would be an attractive alternative. Rocuronium, a new intermediate-acting nondepolarizing neuromuscular blocking agent produces paralysis within 60 seconds, similar to succinylcholine, but has a duration of paralysis of approximately 20 to 30 minutes. If rocuronium-induced paralysis could be chemically reversed within 10 to 15 minutes after the administration of an intubating dose, it may be an appropriate alternative in patients with contraindications to succinylcholine or in patients whom a difficult airway is anticipated. Neostigmine is an anticholinesterase agent which inhibits the hydrolysis of acetylcholine by competing with acetylcholine for attachment to acetylcholinesterase. Inhibition of the breakdown of acetylcholine allows the neurotransmitter to be present in the neuromuscular junction for a longer period of time, so that each molecule can bind repeatedly with the acetylcholine receptor. The purpose of this study is to determine the dose of neostigmine necessary for the early reversal of rocuronium-induced paralysis.

DETAILED DESCRIPTION:
Neuromuscular blocking agents are commonly used to facilitate endotracheal intubation. Succinylcholine, an ultra short-acting, depolarizing neuromuscular blocking agent, is the most commonly used agent for paralysis in this setting because of its rapid onset and short duration of paralysis. In patients with contraindications to succinylcholine or in whom a difficult airway is anticipated, a neuromuscular blocking agent with a pharmacodynamic profile similar to succinylcholine would be an attractive alternative. Rocuronium, a new intermediate-acting nondepolarizing neuromuscular blocking agent produces paralysis within 60 seconds, similar to succinylcholine, but has a duration of paralysis of approximately 20 to 30 minutes. If rocuronium-induced paralysis could be chemically reversed within 10 to 15 minutes after the administration of an intubating dose, it may be an appropriate alternative in patients with contraindications to succinylcholine or in patients whom a difficult airway is anticipated. Neostigmine is an anticholinesterase agent which inhibits the hydrolysis of acetylcholine by competing with acetylcholine for attachment to acetylcholinesterase. Inhibition of the breakdown of acetylcholine allows the neurotransmitter to be present in the neuromuscular junction for a longer period of time, so that each molecule can bind repeatedly with the acetylcholine receptor. The purpose of this study is to determine the dose of neostigmine necessary for the early reversal of rocuronium-induced paralysis.

ELIGIBILITY:
American Society of Anethesiology Class I-III adult patients undergoing elective surgery requiring neuromuscular blockage for endotracheal intubation.

No pre-existing renal or hepatic disease, Myasthenia-Gravis, Eaton-Lambert Disease, pregnancy, concurrent anticonvulsant therapy, history of hypersensitivity to rocuronium, neostigmine, or glycopyrrolate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 1996-09; Study Completion 2000-08

CONTACTS AND LOCATIONS:
Locations (1):
- Warren G. Magnuson Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Martyn JA, White DA, Gronert GA, Jaffe RS, Ward JM. Up-and-down regulation of skeletal muscle acetylcholine receptors. Effects on neuromuscular blockers. Anesthesiology. 1992 May;76(5):822-43. doi: 10.1097/00000542-199205000-00022. PMID 1575351
- [Background] Koide M, Waud BE. Serum potassium concentrations after succinylcholine in patients with renal failure. Anesthesiology. 1972 Feb;36(2):142-5. doi: 10.1097/00000542-197202000-00013. No abstract available. PMID 5059104
- [Background] Mayer M, Doenicke A, Hofmann A, Peter K. Onset and recovery of rocuronium (Org 9426) and vecuronium under enflurane anaesthesia. Br J Anaesth. 1992 Nov;69(5):511-2. doi: 10.1093/bja/69.5.511. PMID 1361356